CLINICAL TRIAL: NCT01670474
Title: Prolonged Hemodialysis Catheter Survival With Copolymer Coating and Rt-PA - PROCOPrt-PA Trial
Brief Title: Prolonged Hemodialysis Catheter Survival With Copolymer Coating and Rt-PA
Acronym: PROCOPrt-PA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier du Centre du Valais (Other)
Responsible Party: Principal Investigator, Pascal Meier MD, Professor, Centre Hospitalier du Centre du Valais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROCOPrt-PA; Cath-a-lysis (Registry Identifier: Dolphin Protect catheter and Actilysis)
Record Dates: First submitted 2012-03-20; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Malfunction; Catheter; Thrombosis; Mechanical Complication of Hemodialysis Catheter
Keywords: Temporary hemodialysis catheters; Non-cuffed hemodialysis catheters; Thrombolysis; rt-PA; Thrombosis; Lifespan; Blood flow rate; Catheter related bacteriemia
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fmDLC and rt-PA (2mg/2mL actilysis) (Experimental): Surface thrombogenicity of film-coated domain structured double lumen catheters (fmDLC) consisting of a novel reactive polyurethane copolymer coating will be assessed by measurement of thrombin-antithrombin (TAT) III complex in vitro after the use of rt-PA (2mg/2mL) in each lumen of the catheter for 45 minutes.
  Each lumen of the thrombosed (dysfunctional) catheter will be locked with the exact volume (luminal volume) of rt-PA (rt-PA (2mg/2mL) actilysis) during 45 min.
  Interventions: Drug: rt-PA (2mg/2mL) actilysis; Drug: rt-PA
- polyDLC and rt-PA (2mg/2mL actilysis) (Active Comparator): The same procedure will be assessed in the polyurethane double lumen catheter (polyDLC)as with the fmDLC. Indeed, surface thrombogenicity of polyDLC will be assessed by measurement of thrombin-antithrombin (TAT) III complex in vitro after the use of rt-PA (2mg/2mL) in each lumen of the catheter for 45 minutes.
  Each lumen of the thrombosed (dysfunctional) catheter will be locked with the exact volume (luminal volume) of rt-PA (rt-PA (2mg/2mL) actilysis) during 45 min.
  Interventions: Drug: rt-PA (2mg/2mL) actilysis; Drug: rt-PA
- siDLC and rt-PA (2mg/2mL actilysis) (Active Comparator): Same procedure as the previous catheters. Surface thrombogenicity of silicone double lumen catheter (siDLC) will be assessed by measurement of thrombin-antithrombin (TAT) III complex in vitro after the use of rt-PA (2mg/2mL) in each lumen of the catheter for 45 minutes.
  Each lumen of the thrombosed (dysfunctional) catheter will be locked with the exact volume (luminal volume) of rt-PA (rt-PA (2mg/2mL) actilysis) during 45 min.
  Interventions: Drug: rt-PA (2mg/2mL) actilysis; Drug: rt-PA

INTERVENTIONS:
Drug: rt-PA (2mg/2mL) actilysis — At the first catheter dysfunction (Qb < 250 ml/min) due to thrombotic event, the patient will receive rt-PA (2mg/2mL Alteplase vial - Cathflo, Boehringer Ingelheim, Ingelheim, Germany). Each lumen of the thrombosed catheter is locked with the exact volume (luminal volume) of rt-PA during 45 min. All catheters analyzed (fmDLC, polyDLC and siDLC) will be locked with the exact volume (luminal volume) of rt-PA during 45 min. Each catheter analyzed will be filled with rt-PA (2mg/2mL) if they are dysfunctional as described above in Arm/Group Descriptions: i.e. fmDLC, polyDLC amd siDLC.
  Other Names: Cathflo, 2mg/2mL (Boehringer Ingelheim, Ingelheim/Germany
Drug: rt-PA — At the first catheter dysfunction (Qb < 250 ml/min) due to thrombotic event, the patient will receive rt-PA (2mg/2mL Alteplase vial - Cathflo, Boehringer Ingelheim, Ingelheim, Germany). Each lumen of the thrombosed catheter is locked with the exact volume (luminal volume) of rt-PA during 45 min. Each catheter analyzed in this study (i.e. fmDLC, polyDLC, siDLC) will be filled with rt-PA (2mg/2mL) if they are dysfunctional as described above in Arm/Group Descriptions.
  Other Names: Cathflo, 2mg/2mL (Boehringer Ingelheim, Ingelheim/Germany)

SUMMARY:
Surface thrombogenicity of standard double lumen catheters (stDLC) and surface modified film-coated domain structured double lumen catheters (fcDLC) consisting of a novel reactive polyurethane copolymer coating showed that in vitro measured surface thrombogenicity was reduced in the modified catheter compared with standard catheter. The clinical investigation revealed that both number of days before catheter removal according to clinical requirements and number of treatments per catheter were significantly higher with the modified catheter as compared with the standard catheter.

Recombinant tissue plasminogen activator (rt-PA) has been used primarily to treat catheter thrombosis. The relatively high cost of rt-PA and its theoretical potential to cause bleeding, as well as the morbidity and mortality associated with catheter malfunction and infection, justify the need for more definitive evidence of the efficacy of rt-PA as a locking solution.

No study aims to evaluate the impact of rt-PA locking in long-term Hemodialysis (HD) uncuffed catheters survival.

DETAILED DESCRIPTION:
The solution instilled into the central venous catheter lumens after each HD session and left in the catheter until the next session (catheter locking solution) is used to prevent thrombosis during the period between HD sessions and may also prevent catheter-related infection. However, evidence supporting the use of various locking solutions to achieve these objectives is limited. Heparin has been the traditional locking solution. Several small studies have assessed whether citrate and heparin are equally efficacious for maintaining catheter patency but the interpretation of the results was limited because the studies had a short follow-up period and included both uncuffed and cuffed central venous catheters.

Thrombosis is a major cause of HD catheter dysfunction, and this problem is rectified by the use of thrombolytic agents, invasive procedures for declotting, or catheter replacement. A thrombus at the tip of the catheter or a fibrin sheath around it may resist local thrombolysis if it is not reached by sufficient concentrations of the drug. Urokinase has traditionally been used as the thrombolytic agent for HD vascular access declotting, and success rates for declotting vary from 55% to 85%. However, successful treatment of occluded central venous catheter (non HD) with recombinant tissue plasminogen activator (rt-PA) or alteplase was recently achieved in more than 1,000 patients with success (function restored in 798 patients [75.0%; 95% CI: 72.3 to 77.6%]). Serious adverse events monitored within 30 days was very rare and efficacy was independent of age, sex, body weight, and catheter type.

ELIGIBILITY:
Inclusion Criteria:

* End-stage kidney disease patients with newly inserted temporary untunnelled dual-lumen catheter
* Naive to study but not naive to catheters (both virgin and non-virgin catheters will be included)
* Expected to use catheter, and to dialyze at study centre, for at least six months
* Frequency of HD 3 times per week
* If indication for catheter was replacement for catheter related infection patients will be eligible after the infection has been treated and the patient has been off antibiotics for 3 HD sessions
* Patient or legal representative able to provide written consent
* Eighteen years of age or older
* Baseline INR ≤ 1.3 (no anticoagulation allowed outside the HD session)
* Baseline platelet count ≥ 60 x 109/L

Exclusion Criteria:

* Use of systemic anticoagulation (if indication for anticoagulation is catheter patency patients may be eligible if the systemic anticoagulation is discontinued and baseline INR is ≤ 1.3)
* Insertion of a new catheter into the femoral vein
* Current use of antibiotics for catheter-related bacteraemia (see inclusion criteria above)
* Major haemorrhage in the prior 4 weeks, defined as bleeding resulting in a drop in haemoglobin of greater than 20 g/L or bleeding requiring transfusion of packed red blood cells with other clinical evidence or suspicion of bleeding
* History of intra-cranial bleed in the prior 4 weeks
* Intra-cranial or intra-spinal neoplasm (current)
* Allergy or intolerance to rt-PA or heparin or its constituents
* Active pericarditis - defined by the presence of a pericardial rub
* Weight ≤ 30 kg or > 130 kg
* Patient pregnant or lactating
* Child bearing potential (i.e. pre-menopausal woman who is not using a reliable method of contraception)
* Major surgery in past 48 hours (CABG, organ biopsy, puncture of non-compressible vessels), or scheduled for major surgery during the study period
* Involvement in another randomized drug trial
* Presence of a fever as defined by a temperature > 38.2°C

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Lifespan patency with the ability to complete HD session in three different UCs using rt-PA locking protocol | 240 days after patients' enrollement
  The ability to achieve blood flow rates of >= 250 mL/min in three different UCs using rt-PA locking protocol if the UCs present a clotting event (complete or partial thrombosis).

SECONDARY OUTCOMES:
The incidence of catheter-related bacteremia after rt-PA use in case of thrombosed UCs | 240 days after patients' enrollement
  The solution instilled into the central venous catheter lumens after each HD session and left in the catheter until the next session (catheter locking solution) is used to prevent thrombosis during the period between HD sessions and may also prevent catheter-related infection.
Economic evaluation of rt-PA in catheter patency after UCs dysfunction | 240 days after patients' enrollement
  An economic evaluation of rt-PA in catheter patency after dysfunction (partial or complete catheter thrombosis) will be conducted.

OTHER OUTCOMES:
Number of patients who complete HD session with short term HD catheters using rt-PA. | 240 days after patients' enrollement
  This analysis aims to see if rt-PA will decrease the incidence of catheter malfunction due to thrombosis in three different UCs of different synthetic material.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Meier, MD, Principal Investigator — CHCVs - RSV - Hôpital du Valais
Locations (1):
- Centre Hospitalier du Centre du Valais (CHCVs), Sion, Valais, Switzerland

REFERENCES:
- [Result] Meier P, Meier R, Turini P, Friolet R, Blanc E. Prolonged catheter survival in patients with acute kidney injury on continuous renal replacement therapy using a less thrombogenic micropatterned polymer modification. Nephrol Dial Transplant. 2011 Feb;26(2):628-35. doi: 10.1093/ndt/gfq449. Epub 2010 Jul 28. PMID 20667989